CLINICAL TRIAL: NCT01195831
Title: Multicentre, Randomized, Investigator-Blinded, Parallel-group Study to Assess the Efficacy and Safety of Xamiol® Gel Compared to Calcipotriol Scalp Solution in Patients With Scalp Psoriasis.
Brief Title: Efficacy and Safety of Xamiol® Gel Compared to Calcipotriol Scalp Solution in Patients With Scalp Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBL 0802 CN
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2015-03

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xamiol® gel (Experimental): Calcipotriol (as hydrate) 50mcg/g plus betamethasone 0.5mg/g (dipropionate)
  Interventions: Drug: Xamiol® gel
- Calcipotriol scalp solution (Active Comparator): Calcipotriol (as hydrate) 50 mcg/ml
  Interventions: Drug: Calcipotriol scalp solution

INTERVENTIONS:
Drug: Xamiol® gel — Once daily application
  Arms: Xamiol® gel
Drug: Calcipotriol scalp solution — Twice daily application
  Arms: Calcipotriol scalp solution

SUMMARY:
The purpose of this study is to compare the clinical efficacy of once daily treatment for 4 weeks with Xamiol® gel (calcipotriol plus betamethasone) with twice daily treatment for 4 weeks with Calcipotriol Scalp Solution in patients with scalp psoriasis.

ELIGIBILITY:
Inclusion Criteria:

Patients of either gender between 18 and 65 years of age.

A clinical diagnosis of scalp psoriasis which is:

* of an investigator's assessment of clinical signs of the scalp at least ≥ 2 in one of the clinical signs, redness, thickness and scaliness, and at least 1 in each of the other two clinical signs, and total score ≥ 4,
* of an extent of 10% or more of the total scalp area,
* of at least moderate severity according the investigator's global assessment.

Clinical signs of psoriasis vulgaris on trunk and/or limbs, or earlier diagnosed with psoriasis vulgaris on trunk and/or limbs.

The patient must provide signed and dated informed consent before any study related activity is carried out.

Exclusion Criteria:

Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis.

Patients with any of the following conditions present on the scalp area: viral lesions, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, acne vilgaris, acne rosacea, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, ulcers and wounds.

Any other inflammatory skin diseases that may confound the evaluation of scalp psoriasis

Systemic treatment with biological therapies (marketed or not marketed), with a possible effect on scalp psoriasis (e.g., alefacept, efalizumab, etanercept, infliximab) within 3 months prior to visit 1 and during the study.

Systemic treatment with all other therapies than biologicals, with a possible effect on scalp psoriasis (e.g., corticosteroids, vitamin D analogues, retinoids, immunosuppressants) within 4 weeks prior to SV2 or during the study.

PUVA therapy within 4 weeks prior to randomisation (visit 1) or during the study.

UVB therapy wthin 2 weeks prior to randomisation (visit 1) or during the study.

Therapies within 2 weeks prior to SV2 and during the study.

* Topical treatment of psoriasis on non scalp psoriasis lesions with potent or very potent (WHO group III-IV) corticosteroids,
* Topical treatment of Immunomodulator, e.g. Tacrolimus,
* Vitamin D analogues (e.g, calcipotriol, tacalcitol, calcitriol),
* Any topical treatment of the scalp (except for non-steroid medicated shampoos and emollients,
* Other types of psoriasis treatment, e.g. Chinese medicine, processed Chinese medicine, or hot spring, etc.

Planned initiation of, or changes to concomitant medication that could affect scalp psoriasis (e.g., beta blockers, anti-malaria drugs, lithium) during the study.

Known or suspected hypersensitivity to component(s) of the Investigational Products.

Known or suspected abnormality of the calcium homeostasis.

Known or suspected severe renal insufficiency or severe hepatic disorders, or severe heart disease.

Clinical signs or symptoms of Cushing's disease or Addison's disease.

Planned extensive exposure to sun (e.g. when working outdoors) during the study, which may affect scalp psoriasis.

Females who are pregnant, or of child-bearing potential and wish to become pregnant during the study, or who are breast-feeding.

Females of child-bearing potential with a positive serum or urine pregnancy test at SV2.

Any clinically significant abnormality following review of screening laboratory tests (blood and urine samples), physical examination or blood pressure/heart rate measurement performed at SV2.

Participation in any other interventional clinical trial within 4 weeks prior to randomisation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Xu, Professor, Principal Investigator — China
Locations (9):
- China (9):
  - Bei Jing Hospital Affiliated Ministry of Health, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital Affiliated to Peking University, Beijing
  - Southwest Hospital Affiliated to Third Military Medical University, Chongqing
  - Second Hospital Affiliated to Medical College of Zhe Jiang University, Hangzhou
  - Chinese Academy of Medical Sciences & Peking Union Medical College, Institute of Dermatology, Nanjing, Nanjing
  - Changhai Hospital Affiliated to Second Military Medical University, Shanghai
  - Huashan Hospital Affiliated to Fu Dan University, Shanghai
  - Xi Jing Hospital Affiliated to Fourth Military Medical University Xi Jing Hospital, Xi'an

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study period was 17 September 2010 (date of the first enrolment) to 01 March 2011 (date of last patient out)
Period: Overall Study
Arm/Group | Xamiol® Gel | Calcipotriol Scalp Solution
Started | 120 | 124
Completed | 112 | 114
Not Completed | 8 | 10
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 4 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xamiol® Gel | Calcipotriol Scalp Solution | Total
Number analyzed (Participants) | 120 | 124 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.87 (13.145) | 38.73 (11.869) | 39.29 (12.500)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 55 | 102
  Male | 73 | 69 | 142
Region of Enrollment [Number; unit: participants]
  China | 120 | 124 | 244

OUTCOME MEASURES:

1. Primary Outcome: Patients With "Controlled Disease" in Terms of "Clear" or "Minimal" According to Investigator's Global Assessment of Disease Severity at Week 4.
Description: Investigators made a global assessment of the disease severity by use of a 6-point scale (Clear, Minimal, Mild, Moderate, Severe and Very Severe). Patients with disease severity classified as Clear or Minimal disease after the treatment period (week 4) were rated as having Controlled disease.
Time Frame: 4 weeks
Measure: Number; unit: percentage of parcipitants
Arm/Group | Xamiol® Gel | Calcipotriol Scalp Solution
Number analyzed (Participants) | 120 | 124
percentage of parcipitants | 87.5 | 50.8

2. Secondary Outcome: Patients With "Controlled Disease" in Terms of "Clear" or "Minimal" According to Investigator's Global Assessment of Disease Severity at Week 2
Description: Investigators made a global assessment of the disease severity by use of a 6-point scale (Clear, Minimal, Mild, Moderate, Severe and Very Severe). Patients with disease severity classified as Clear or Minimal disease at week 2 were rated as having Controlled disease.
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Xamiol® Gel | Calcipotriol Scalp Solution
Number analyzed (Participants) | 120 | 124
percentage of participants | 80.8 | 25.8

3. Secondary Outcome: Patients With "Controlled Disease" in Terms of "Clear" or "Very Mild" According to Patient's Global Assessment of Disease Severity at Week 2.
Description: Patients made a global assessment of the disease severity by use of a 5-point scale (Clear, Very Mild, Mild, Moderate, Severe). Patients classifying their disease as Clear or Very Mild at week 2 were rated as having Controlled disease. This assessment was made prior to the investigator's assessments.
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Xamiol® Gel | Calcipotriol Scalp Solution
Number analyzed (Participants) | 120 | 124
percentage of participants | 79.2 | 37.1

4. Secondary Outcome: Patients With "Controlled Disease" in Term of "Clear" or "Very Mild" According to Patient's Global Assessment of Disease Severity at Week 4.
Description: Patients made a global assessment of the disease severity by use of a 5-point scale (Clear, Very Mild, Mild, Moderate, Severe). Patients classifying their disease as Clear or Very Mild at week 4 were rated as having Controlled disease. This assessment was made prior to the investigator's assessments.
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Xamiol® Gel | Calcipotriol Scalp Solution
Number analyzed (Participants) | 120 | 124
percentage of participants | 90.8 | 60.5

5. Secondary Outcome: Patients With Success (Total Sign Score ≤1) at Week 4
Description: Investigators assessed scalp psoriasis lesions in terms of three clinical signs: redness, thickness and scaliness. For each clinical sign a single score, reflecting the average severity of all lesions on the scalp, was derived according to a 5-point scale ranging from 0 to 4 (0= best;4= worst). The sum of the three individual scores (redness, thickness and scaliness) constituted a Total Sign Score of the scalp ranging from 0 to 12 (0= best;12= worst). Patients with a Total sign score of 0 or 1 at week 4 achieved "Success".
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Xamiol® Gel | Calcipotriol Scalp Solution
Number analyzed (Participants) | 120 | 124
percentage of participants | 64.2 | 25.8

6. Secondary Outcome: For Each Clinical Sign (Redness, Thickness, Scaliness), the Percentage of Patients With Success (Clinical Score=0) at Week 4
Time Frame: 4 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Patients With Success (Patient's Itching Score=None) at Week 4
Time Frame: 4 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Evaluation of the Quality of Life
Time Frame: Baseline to weeks 2 and 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The Number of participants at risk is based on the number of participants included in the safety analysis set, i.e. all randomized patients who had at least one dose of medication, and had at least one post-baseline safety assessment (118 out of 120 patients in Xamiol® gel group and all (124) patients in Calcipotriol scalp solution group)
Arm/Group | Xamiol® Gel | Calcipotriol Scalp Solution
Serious Adverse Events (participants affected / at risk) | 2/118 | 0/124
Other Adverse Events (participants affected / at risk) | 15/118 | 36/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xamiol® Gel (N=118) | Calcipotriol Scalp Solution (N=124)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xamiol® Gel (N=118) | Calcipotriol Scalp Solution (N=124)
Application site pain (General disorders) | 3 | 14
Application site warmth (General disorders) | 1 | 13
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 11 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The company acknowledges the investigators' right to publish the results of the trial. The company retains the right to have any publication submitted to the company for review at least 30 days prior to the proposed submission or presentation date. Investigators must undertake not to submit any part of their individual data for publication without prior consent of LEO.